CLINICAL TRIAL: NCT06179875
Title: An Open-label Study for Participants Who Are Non-responders at the End of Treatment Assessment on the VRDN-001-101 and VRDN-001-301 Pivotal Studies
Brief Title: An Open-label Study (OLE) for Non-responders of VRDN-001-101 and VRDN-001-301
Acronym: OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Viridian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRDN-001-302
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Eye Disease
Keywords: Graves; Thyroid-Associated Ophthalmopathy; Thyroid Eye Disease; Dysthyroid Ophthalmopathy; Graves Eye Disease; Graves Orbitopathy; Myopathic Ophthalmopathy; Congestive Ophthalmopathy; Edematous Ophthalmopathy; Infiltrative Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methods; Therapeutics

STUDY DESIGN:
Intervention Model Description: Single treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VRDN-001 10 mg/kg (Experimental): 5 infusions of VRDN-001 10 mg/kg
  Interventions: Drug: Intervention/Treatment

INTERVENTIONS:
Drug: Intervention/Treatment — VRDN-001 10 mg/kg (5 infusions of VRDN-001 10 mg/kg)

SUMMARY:
The investigational drug, VRDN-001, is a monoclonal antibody that inhibits the activity of a cell surface receptor called insulin-like growth factor-1 receptor (IGF-1R). Inhibition of IGF-1R may help to reduce the inflammation and associated tissue swelling that occurs in patients with thyroid eye disease (TED). The primary objectives of this clinical trial are to provide open-label access to VRDN-001 for participants who were previously non-responders at 3 weeks post the fifth IV infusion (i.e., 15 weeks) in the VRDN-001-101 (THRIVE) and VRDN-001-301 (THRIVE-2) pivotal studies and assess the safety and efficacy of VRDN-001 in participants who were previously treated with VRDN-001 or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Be able to understand the study procedures and the risks involved and be willing to provide written informed consent before the first study-related activity
2. Have completed at least 5 IV infusions and assessments required to determine proptosis responder status 3 weeks post the fifth IV infusion (i.e., Week 15) as defined in either the VRDN-001-101 or VRDN-001-301 pivotal studies
3. Been a participant in either the VRDN-001-101 or VRDN-001-301 studies and found to be a non-responder as defined within the VRDN-001-101 or VRDN-001-301 study
4. Not require immediate surgical ophthalmological or orbital surgery in the study eye for any reason
5. Must agree to use highly effective contraception as specified in the protocol
6. Female TED participants must have a negative urine pregnancy test at screening
7. Be willing and able to comply with all the requirements of the protocol for the entire duration of the study

Key Exclusion Criteria:

Participants must not:

1. Have received prior treatment with another anti-IGF-1R agent
2. Have received systemic corticosteroids for any condition, including TED, or selenium within 2 weeks prior to first dose
3. Have received other immunosuppressive drugs or another investigational agent for any condition, including TED (other than VRDN-001 or placebo associated with the VRDN-001-101 or VRDN-001-301 pivotal studies), or any other therapy for TED, within 8 weeks prior to first dose
4. Have received radioactive iodine (RAI) treatment within 8 weeks prior to first dose
5. Have had previous orbital irradiation or decompression surgery involving excision of fat for TED to the study eye's orbit
6. Have abnormal hearing test before first dose. Have a history of ear conditions considered significant by study doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Proptosis Responder Rate in the most proptotic eye | Week 15
  Proptosis Responder Rate in the most proptotic eye (i.e., reduction of proptosis of ≥ 2 mm from baseline [without a corresponding increase of ≥ 2 mm in the other eye]) as measured by exophthalmometer

SECONDARY OUTCOMES:
Change from Baseline in proptosis in the most proptotic eye | Week 15
  Change from Baseline in proptosis in the most proptotic eye as measured by exophthalmometer
Proptosis Responder Rate in the most proptotic eye | Week 15
  Proptosis Responder Rate in the most proptotic eye as measured by MRI/CT
Change from baseline in proptosis in the most proptotic eye | Week 15
  Change from baseline in proptosis in the most proptotic eye as measured by MRI/CT
Clinical Activity Responder Rate in the most proptotic eye | Week 15
  Clinical Activity Responder Rate in the most proptotic eye as measured by exophthalmometer
Overall Responder Rate in the most proptotic eye | Week 15
  Overall Responder Rate in the most proptotic eye as measured by exophthalmometer and Clinical Activity Responder Rate in the most proptotic eye as measured by exophthalmometer
Diplopia Responder Rate | Week 15
  Diplopia Responder Rate (i.e., reduction in Gorman Subjective Diplopia Score of ≥1 from baseline for participants with baseline Gorman Subjective Diplopia Score >0).
Diplopia Resolution Rate | Week 15
  Diplopia Resolution Rate (i.e., reduction in Gorman Subjective Diplopia Score to 0 from baseline for participants with baseline Gorman Subjective Diplopia Score >0).

CONTACTS AND LOCATIONS:
Locations (45):
- United States (18):
  - Advancing Research International, LLC, Los Angeles, California
  - USC Eye Institute, Los Angeles, California
  - Advancing Research International, LLC, Newport Beach, California
  - Stanford Byers Eye Institute, Palo Alto, California
  - Cockerham Eye Consultants, PC, San Diego, California
  - University of Miami Miller School of Medicine, Bascom Palmer Eye Institute, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Vision Medical Research, Oak Lawn, Illinois
  - Ophthalmic Consultants of Boston, East Weymouth, Massachusetts
  - Kahana Oculoplastic & Orbital Surgery, Livonia, Michigan
  - Ophthalmic Plastic, Reconstructive, Orbital and Cosmetic Surgery, Las Vegas, Nevada
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - The Center for Eye and Facial Plastic Surgery, Somerset, New Jersey
  - Hospital of the University of Pennsylvania Perleman Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Neuro-Eye Clinical Trials, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington
- France (3):
  - CHU Angers, Angers, France
  - Centre Hospitalier Universitaire de Montpellier Hopital Lapeyronie, Montpellier, Hérault
  - Centre Hospitalier Universitaire De Nantes G.R. Laenne, Saint-Herblain, Loire-Atlantique
- Germany (5):
  - Universitatmedizin Gottingen, Göttingen, Lower Saxony
  - Charite - Universitatsmedizin Berlin KoR, Campus Virchow Klinikum, Klinik tor Augenheilkunde, Berlin
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Essen AoR - Klinik fur Augenheilkunde, Essen
  - University Medical Center Freiburg, Freiburg im Breisgau
- Amsterdam UMC, Amsterdam, Netherlands
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Bialystok
  - Optimum Profesorskie Centrum Okulistyki, Gdansk, Gdansk
  - Centrum Medyczne Pulawska, Piaseczno, Piaseczno
  - Centrum Medyczne Piasta, Wałbrzych, Piasta
- Spain (5):
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Arruzafa. Servicio de Oftalmologia, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Miguel Servel, Zaragoza
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Tip Fakultesi, Ankara, Ankara
  - Gazi University Medical Faculty Hospital, Ankara, Ankara
  - Akdeniz University Medical Faculty Hospital, Antalya, Antalya
  - Marmara University Faculty of Medicine, Istanbul, Istanbul
- United Kingdom (5):
  - Imperial College Healthcare NHS Trust Western Eye Hospital, London, London
  - Guy's and St. Thomas Trust, London, London
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich, London
  - University Hospital Bristol and Weston NHS Foundation Trust- Bristol Eye Hospital, Bristol
  - Newcastle Eye Centre, Newcastle